CLINICAL TRIAL: NCT06096922
Title: Frailty Assessment Tool for Patients Undergoing Cardiac Surgery Based on Artificial Intelligence Multimodal Non-contact Monitoring.
Brief Title: AI-based Frailty Assessment Tool for Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-GSP-RC-10
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Frailty
Keywords: Frailty; Cardiac surgery; Artificial intelligence; Non-contact monitoring
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AI frailty index establishment group: Individuals who undergo elective cardiac surgury
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The main purpose of this study is to establish a frailty automatic evaluation index "AI frailty index" based on artificial intelligence multi-modal non-contact monitoring information analysis. At the same time, the study will explore the correlation between ' AI weakness index ' and perioperative and long-term prognosis and quality of life.

DETAILED DESCRIPTION:
This is a prospective cohort study. Patients who undergoes elective cardiac surgery will be enrolled. We collect frailty scales, clinical information and multi-modal, non-contact monitoring information during hospitalization. One-year follow-up will be done. The non-contact monitoring information are used to predict the frailty scales to establish and validate an AI-based frailty assessment model "AI frailty index". The AI frailty index will be further used to predict perioperative and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Age ≤ 18 years
* The clinical situation is unstable, such as frequent occurrence of coronary ischemia events, unstable heart failure, or acute events leading to severe discomfort symptoms or changes in vital signs
* Unable to cooperate in completing research data collection due to severe neurological and psychiatric abnormalities or other reasons
* Duration of postoperative ventilation > 48 hours or inability to obtain scale data on the first day after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 18 years or older, undergoing elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
One-dimensional matrix vector composed of five frailty scale results | Before and after surgery, up to 2 weeks
  Consisting of five frailty scales: Edmonton frailty scale, FRAIL frailty scale, Fried frailty scale, Clinical frailty scale, and SPPB

SECONDARY OUTCOMES:
30-day adverse events | 30 days post operative
  Including death, readmission, stroke, myocardial infarction, renal insufficiency or renal failure, dialysis, atrial fibrillation, peripheral vascular embolism, bleeding events, heart failure
1-year adverse events | 1 year post operative
  Including death, readmission, stroke, myocardial infarction, renal insufficiency or renal failure, dialysis, atrial fibrillation, peripheral vascular embolism, bleeding events, heart failure
EQ-5D score | 1 year post operative
  The score of EQ-5D questionnaire
QOR-15 score | 1 year post operative
  The score of QOR-15 questionnaire
Edmonton frailty scale score | 1 year post operative
  The Edmonton frailty scale consists of 11 items for a composite score of 0 to 17, and higher scores mean a worse outcome.
FRAIL frailty scale score | 1 year post operative
  The FRAIL frailty scale consists of 5 items, with 3 of 5 required to diagnose frailty.
Fried frailty scale score | 1 year post operative
  The Fried frailty scale consists of 5 items, with 3 of 5 required to diagnose frailty.
Clinical frailty scale score | 1 year post operative
  The Clinical frailty scale is scored 1 to 9 based on a semiquantitative evaluation of the patient's symptoms, mobility, inactivity, exhaustion, and disability for basic activities of daily living and instrumental activities of daily living, and higher scores mean a worse outcome.
Short Physical Performance Battery scale score | 1 year post operative
  The Short Physical Performance Battery scale consists of 3 physical tests, with each scored 0 to 4 for a composite score of 0 to 12, and higher scores mean a better outcome.
Perioperative adverse events | From surgery to discharge, up to 7 days
  Including all cause death, stroke, renal insufficiency, deep sternal wound infection, and reoperation
Area under receiver operating curve (AUC) | At the end of follow-up (1 mouth)
  Area under receiver operating curve of algorithm in predicting frailty scales and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No